CLINICAL TRIAL: NCT03233126
Title: A Phase 3 Open-Label Trial to Assess the Efficacy and Safety of KRN23 in Pediatric Patients With X-linked Hypophosphatemic Rickets/Osteomalacia and a Postmarketing Study of KRN23 Switched From the Phase 3 Trial
Brief Title: A Study of KRN23 in Pediatric Patients With X-linked Hypophosphatemic Rickets/Osteomalacia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN23-003
Record Dates: First submitted 2017-07-11; First posted 2017-07-28 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: X-linked Hypophosphatemic Rickets/Osteomalacia
MeSH Terms: conditions — Familial Hypophosphatemic Rickets; Osteomalacia | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KRN23 (Experimental): Subjects will receive subcutaneous injections of KRN23 every 2 weeks from Week 0 through Week 128
  Interventions: Drug: KRN23

INTERVENTIONS:
Drug: KRN23 — Subjects will receive subcutaneous injections of KRN23 every 2 weeks from Week 0 through Week 86

SUMMARY:
Before switching to the post-marketing study:

To evaluate the efficacy and safety of KRN23 administered subcutaneously once every 2 weeks in children with X-linked hypophosphatemic rickets/osteomalacia(XLH).

After switching to the post-marketing study:

To evaluate the safety and efficacy of KRN23, which is switched from the investigational product to the post-marketing study drug, at the approved dose and dosing regimen in subjects who continue treatment

ELIGIBILITY:
Inclusion Criteria:

1）Personally submitted voluntary written informed consent by a legally authorized representative.If appropriate, written or verbal assent to participate in the study should be obtained from patients.

2) Aged ≥ 1 and ≤12 years 3）Patients who have open growth plate 4）Willing to perform a self-administration of KRN23 and available to perform a self-administration 5）Diagnosis of XLH, and meeting any of the followings;

1. phosphate-regulating gene with homologies to endopeptidases on the X chromosome(PHEX) mutation in either the patient or in a directly related family member with appropriate X-linked inheritance
2. Serum intact FGF23 level at screening ≥ 30 pg/mL 6） Finding evidence of rickets or clinical symptoms 7）Meeting all of following criteria for laboratory test related to XLH;

a）Serum P: < 3.0 mg/dL b）Serum Cr: Within the age-adjusted normal limits c）Serum 25(OH)D: ≥ 16 ng/mL 8） For female patients who have reached menarche with child bearing potential; a negative urine pregnancy test at screening 9）For female patients with child baring potential, or male patients with reproductive capacity; willingness to use an acceptable method of contraception while participating in the study 10） Willingness to provide access to prior medical records to determine eligibility including data on imaging tests, blood chemistry, diagnosis, medication, and surgical history 11） Willingness and ability to cooperatively complete all study procedures, adhere to the visit schedule and follow the investigator's instructions, as considered by the investigator or subinvestigator

Exclusion Criteria:

1）Height percentile > 50% based on age-adjusted Japanese norms at screening 2）Use of aluminum hydroxide antacids, systemic corticosteroids, acetazolamide, and thiazides within 7 days prior to screening 3）Current or prior use of leuprorelin, triptorelin, goserelin, or other drugs known to delay puberty 4）Use of growth hormone therapy within 12 months before screening 5）Use of medication to suppress parathyroid hormone within 60 days prior to screening 6）Serum calcium levels outside the age-adjusted normal limits 7）Intact parathyroid hormone(iPTH) levels ≥ 163 pg/mL 8）Presence of nephrocalcinosis on renal ultrasound grade 4 based on the following scale: 0 = Normal

1. = Faint hyperechogenic rim around the medullary pyramids
2. = More intense echogenic rim with echoes faintly filling the entire pyramid
3. = Uniformly intense echoes throughout the pyramid
4. = Stone formation: solitary focus of echoes at the tip of the pyramid 9）Planned or recommended orthopedic surgery 10）Blood or blood product transfusion within 60 days prior to screening 11）History of malignancy within 5 years prior to registration 12）History of being positive for human immunodeficiency virus antibody, hepatitis B antigen and/or hepatitis C virus antibody 13）Predisposition to infection, or history of recurrent infection or known immunodeficiency 14）Use of any investigational product or investigational medical device within 4 months prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments 15）Receiving investigational agent in the UX023-CL301 study 16）Use of a therapeutic monoclonal antibody other than KRN23 within 90 days prior to screening 17）History of allergic or anaphylactic reactions to KRN23, any of the KRN23 ingredients, or any other monoclonal antibodies 18）Anyone otherwise considered unsuitable participation in the study by the investigator or subinvestigator

Subjects eligible for enrollment in the post-marketing clinical study must meet both of the following criteria:

1) Personally submitted voluntary written informed consent to participate in the postmarketing clinical study by a legally authorized representative. If appropriate, written or verbal assent to participate in the post-marketing clinical study should be obtained from subjects.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Number of subjects for each adverse events | up to week 128
Percentage of subjects for each adverse events | up to week 128

SECONDARY OUTCOMES:
Effect to body temperature | up to week 128
Effect to pulse rate | up to week 128
Effect to respiratory rate | up to week 128
Effect to blood pressure | up to week 128
Effect to 12-Lead Electrocardiogram | up to week 128
Effect to Renal Ultrasound | up to week 128
Effect to Echocardiogram | up to week 128
Serum phosphorus concentration at each test time point | up to week 128
1,25(OH)2D at each test time point | up to week 128
Alkaline phosphatase at each test time point | up to week 128
Urine phosphorus at each test time point | up to week 128
Tubular reabsorption of phosphate at each test time point | up to week 128
TmP/GFR at each test time point | up to week 128
Change from baseline in serum phosphorus | up to week 128
Change from baseline in 1,25(OH)2D | up to week 128
Change from baseline in alkaline phosphatase | up to week 128
Change from baseline in urine phosphorus | up to week 128
Change from baseline in tubular reabsorption of phosphate | up to week 128
Change from baseline in TmP/GFR | up to week 128
Improvement in Radiographic Global Impression of Change(RGI-C) global score | up to week 128
Change from baseline on Rickets Severity Score (RSS) total score | up to week 128
Change from baseline in the Six Minute Walk Test | up to week 128
Change in height-for-age z-scores from baseline | up to week 128
Serum KRN23 concentration | up to week 128
Anti-KRN23 antibody | up to week 128

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Kanagawa Prefectural Hospital Organization Kanagawa Children's Medical Center, Yokohama, Kanagwa
  - Osaka Hospital, Japan Community Healthcare Organization (JCHO), Osaka, Osaka
  - National University Corporation Osaka University Hospital, Suita, Osaka
  - Okayama Saiseikai General Hospital Outpatient Center, Okayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kubota T, Namba N, Tanaka H, Muroya K, Imanishi Y, Takeuchi Y, Kanematsu M, Sun W, Seino Y, Ozono K. Self-Administration of Burosumab in Children and Adults with X-Linked Hypophosphataemia in Two Open-Label, Single-Arm Clinical Studies. Adv Ther. 2023 Apr;40(4):1530-1545. doi: 10.1007/s12325-022-02412-x. Epub 2023 Jan 31. PMID 36719566